CLINICAL TRIAL: NCT04571463
Title: Etyyliglukuronidin Esiintyminen Virtsassa äitiysneuvola- ja äitiyspoliklinikkakäyntien yhteydessä HUS:n ja PHHYKY:n Alueella
Brief Title: Ethyl Glucuronide in Urine Samples of Pregnant Women Within the HUS ja PHHYKY Area
Status: Completed | Type: Observational
Sponsor: Hanna Kahila (Other)
Collaborators: Finnish Pediatric Neurology Association (Unknown); Finnish Foundation for Alcohol Studies (Other); Päijänne Tavastia Central Hospital (Other); Helsinki University Central Hospital (Other); Seinajoki Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Hanna Kahila, Senior Ward Physician, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Other Study IDs: HUS/483/2020
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HUCS A: Mothers visiting the prenatal care units within the Helsinki area.
- HUCS HAL: Mothers visiting the prenatal care units dedicated for the alcohol and drug abusing mothers within the Helsinki area.
- PHHYKY A: Mothers visiting the prenatal care units within the Lahti area.
- PHHYKY HALSO: Mothers visiting the prenatal care units dedicated for the alcohol and drug abusing mothers within the Lahti area.

SUMMARY:
In order to find how many women continue using alcohol during their pregnancies the plan is to anonymously test routine urine samples collected during pregnancies for ethylglucuronide (ETG), a metabolite of ethanol that is detectable in urine up to several days after alcohol consumptions. Altogether 600 samples are taken in the prenatal care units and the prenatal care units dedicated for the alcohol and drug abusing mothers both in the Helsinki and Lahti areas. Test results are used to estimate and compare the prevalence of severe maternal drinking in the different populations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population for the ethylglucuronide (EtG) testing consists of the visitors in the HYKS, PHHYKY and the cities of Helsinki and Lahti prenatal care units, as well as the HYKS and PHHKYKY prenatal care units dedicated for the alcohol and drug abusing mothers (HAL- / HALSO-poliklinikka).
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
EtG | Day 1
  The routine urine samples from the visitors are tested for ethyl glucuronide using dip sticks with 300ng cut off. Positve finds are confirmed in a laboratory.

SECONDARY OUTCOMES:
Nicotine | Day 1
  The positive EtG urine samples and random negative urine samples from the visitors are tested for nicotine using dip sticks.
Cannabis | Day 1
  The positive EtG urine samples and random negative urine samples from the visitors are tested for cannabis using dip sticks.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Kahila, MD, Principal Investigator — HUCS
Locations (4):
- Finland (4):
  - HALSO-poliklinikka, Lahti, Paijat-Hame Region
  - Äitiyspoliklinikka/neuvola, Lahti, Paijat-Hame Region
  - HAL-poliklinikka, Helsinki, Uusimaa
  - Äitiyspoliklinikka/neuvola, Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: Yes
All collected anonymized IPD and the modeling source code will be shared.
Supporting Information: ICF, Analytic Code
Time Frame: 6 months after the publication
Access Criteria: Scientific study, policy making

REFERENCES:
- [Derived] Jolma M, Koivu-Jolma M, Niemela O, Autti-Ramo I, Kahila H. Rapid urine screening for ethyl glucuronide from pregnant women as a tool for detecting prenatal alcohol exposure. BMC Pregnancy Childbirth. 2023 Jun 22;23(1):464. doi: 10.1186/s12884-023-05789-x. PMID 37349673